CLINICAL TRIAL: NCT07320040
Title: Evaluation of Emotion-related Salivary Molecular Biomarkers Following Olfactory Stimuli
Brief Title: Evaluation of Emotion-related Salivary Molecular Biomarkers
Acronym: EMJOY
Status: Recruiting | Type: Observational
Sponsor: Sys2Diag (Other Government)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Principal Investigator, Laurence MOLINA, Project Manager, Sys2Diag
Other Study IDs: 2022-A02008-35; 22.03698.000189 (Other: Comité de protection des personnes (French Ethics committee))
Record Dates: First submitted 2025-12-19; First posted 2026-01-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Emotion
Keywords: Biomarkers; Stimuli; Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bras S Fragrance then placebo: Subjects will be subjected successively to fragrance and placebo stimulation.
  Interventions: Other: Identication and measurement of a molecular biomarkers signature
- Bras P Placebo then fragrance: Subjects will be subjected successively to placebo and fragrance stimulation.
  Interventions: Other: Identication and measurement of a molecular biomarkers signature

INTERVENTIONS:
Other: Identication and measurement of a molecular biomarkers signature — Levels of the biomarkers of interest (DHEA, pg/mL; Oxytocin, pg/mL; Cortisol, pg/mL; Alpha Amylase, U/mL) will be measured in the saliva of participating subjects by enzymatic assay methods or ELISA-type methods performed using commercial kits.

SUMMARY:
Recent studies show that emotional states can be discriminated by physiological responses. This physiological regulation results from the action of enzymes and hormones that represent the activity of the autonomic nervous system. The measurement of specific biomarkers, using non-invasive biological tests in saliva, would therefore provide physiological data on an individual's emotional state in response to stimuli, particularly olfactory stimuli.

DETAILED DESCRIPTION:
Recent studies show that emotional states (positive and negative) can be discriminated by physiological responses. This physiological regulation stems from the action of enzymes and hormones that represent the activity of the autonomic nervous system. The measurement of specific biomarkers (enzymes, hormones), using non-invasive biological tests in saliva, would therefore provide physiological data on an individual's emotional state (Giacomello et al. 2020) in response to stimuli, particularly olfactory stimuli.

The aim of the proposed research is to identify and measure a signature of molecular biomarkers in saliva, linked to emotions following one or more olfactory stimuli (e.g. cortisol and alpha-amylase concentration increase after stimulation).

ELIGIBILITY:
Inclusion Criteria:

* Subject willing to follow study procedures
* Subject able to understand the purpose, nature and methodology of the study
* Subject has signed informed consent form
* Subjects between 18 and 60 years of age.

Exclusion Criteria:

* Subjects deprived of liberty, protected adults, vulnerable persons or minors
* Subjects with a proven or suspected chronic infectious disease that could entail a risk of contamination during sample handling (laboratories not equipped to handle this type of sample)
* Rejection to sign the consent form.

Non specific inclusion criteria:

* Pregnant or breastfeeding women
* Subjects presenting anosmia during the last 15 days
* Subjects presenting symptoms and signs of active oral inflammation, advanced periodontitis or severe gingivitis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population for this study will consist of healthy volunteers who meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2027-06-14 (Estimated)

PRIMARY OUTCOMES:
Evaluate variations | 1 year
  Evaluate variations in several molecular biomarkers in saliva following fragrance stimulus/stimuli that may be linked to an emotionnal response (positive or negative).

SECONDARY OUTCOMES:
Identify a molecular biomarker signature | 2 years
  Identify a molecular biomarker signature in saliva following fragrance stimulus or stimuli.
Evaluate basal values of biomarkers | 3 years
  Evaluate basal values of biomarkers composing the signature under normal, unstimulated conditions (intra-individual, inter-individual variations, circadian rhythm, age, gender...).
Evaluate signature dynamics | 1 year
  Evaluate signature dynamics after stimulation
Establish correlations between biomarker signatures and emotion ratings | 3 years
  Establish correlations between biomarker signatures and emotion ratings based on other criteria, such as questionnaires.
Compare biomarker signatures | 2 years
  Compare biomarker signatures in response to different fragrance stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence MOLINA, Phd, Principal Investigator — Sys2Diag
Locations (1):
- SYS2DIAG - UMR9005 CNRS/ALCEN, Montpellier, 34184, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giacomello G, Scholten A, Parr MK. Current methods for stress marker detection in saliva. J Pharm Biomed Anal. 2020 Nov 30;191:113604. doi: 10.1016/j.jpba.2020.113604. Epub 2020 Sep 6. PMID 32957066